CLINICAL TRIAL: NCT01816607
Title: Functional MRI of Hypoxia-mediated Rectal Cancer Aggressiveness
Acronym: OxyTarget
Status: Completed | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Collaborators: Oslo University Hospital (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Kathrine Røe Redalen, Senior scientist, University Hospital, Akershus
Other Study IDs: REK-2013/152; REK-2013/152 (Other Grant/Funding Number: HSØ_2013002)
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Rectal Diseases; Rectal Neoplasms; Gastrointestinal Diseases; Gastrointestinal Neoplasms
Keywords: Magnetic Resonance Imaging; Magnetic Resonance Imaging, Functional
MeSH Terms: conditions — Rectal Diseases; Rectal Neoplasms; Gastrointestinal Diseases; Gastrointestinal Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, rectal cancer tissue, normal tissue, lymph nodes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rectal cancer
  Interventions: Procedure: new functional magnetic resonance imaging (MRI) protocols

INTERVENTIONS:
Procedure: new functional magnetic resonance imaging (MRI) protocols — diffusion-weighted MRI, dynamic-contrast enhanced MRI, MR spectroscopy, blood-level oxygen dependent (BOLD) MRI

SUMMARY:
The purpose of this study is to establish a reliable method for detection of rectal cancer patients with aggressive tumor at risk of metastatic disease and death by functional MRI.

ELIGIBILITY:
Inclusion Criteria:

* The patient is willing and able to give full written consent according to the protocol approved by the Regional Ethics Committee.
* The patient has confirmed rectal cancer diagnosis and is scheduled to radical surgery alone or preoperative CRT followed by surgery.
* The patient is ≥ 18 years.
* The patient has no prior rectal cancer treatment.
* The patient has adequate renal function: creatinine clearance ≥ 60 ml/minute.
* The patient has signed the written informed consent according to the protocol approved by the Regional Ethics Committee.

Exclusion Criteria:

* The patient has contraindication to MRI or MRI contrast agent according to clinical practice.
* The patient wants to withdraw for any reason during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rectal cancer patients referred to radical surgery, with or without preoperative chemoradiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2013-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Presence of metastatic disease 5 years after rectal cancer treatment | five years

SECONDARY OUTCOMES:
Histomorphological response to preoperative chemoradiotherapy | 8 weeks

OTHER OUTCOMES:
Detection of regional malignant lymph nodes at time of diagnosis | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathrine Røe Redalen, PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lørenskog, Akershus, Norway

REFERENCES:
- [Result] Bousquet PA, Meltzer S, Sonstevold L, Esbensen Y, Dueland S, Flatmark K, Sitter B, Bathen TF, Seierstad T, Redalen KR, Eide L, Ree AH. Markers of Mitochondrial Metabolism in Tumor Hypoxia, Systemic Inflammation, and Adverse Outcome of Rectal Cancer. Transl Oncol. 2019 Jan;12(1):76-83. doi: 10.1016/j.tranon.2018.09.010. Epub 2018 Sep 29. PMID 30273860
- [Result] Grovik E, Redalen KR, Storas TH, Negard A, Holmedal SH, Ree AH, Meltzer S, Bjornerud A, Gjesdal KI. Dynamic multi-echo DCE- and DSC-MRI in rectal cancer: Low primary tumor Ktrans and DeltaR2* peak are significantly associated with lymph node metastasis. J Magn Reson Imaging. 2017 Jul;46(1):194-206. doi: 10.1002/jmri.25566. Epub 2016 Dec 21. PMID 28001320
- [Derived] Bakke KM, Bjornetro T, Bousquet PA, Sanabria AM, Meltzer S, Luders T, Troseid AS, Stang E, Negard A, Froyen EA, Lunder AK, Lyckander LG, Aass HCD, Redalen KR, Ree AH. Dissemination of Mitochondrial DNA Variants: Looking at the 'Bigger' Picture of the Tumour Microenvironment in Rectal Cancer Patients. J Extracell Biol. 2025 Oct 30;4(11):e70097. doi: 10.1002/jex2.70097. eCollection 2025 Nov. PMID 41179924
- [Derived] Bjornetro T, Bousquet PA, Redalen KR, Troseid AS, Luders T, Stang E, Sanabria AM, Johansen C, Fuglestad AJ, Kersten C, Meltzer S, Ree AH. Next-generation sequencing reveals mitogenome diversity in plasma extracellular vesicles from colorectal cancer patients. BMC Cancer. 2023 Jul 12;23(1):650. doi: 10.1186/s12885-023-11092-x. PMID 37438741
- [Derived] Bousquet PA, Meltzer S, Fuglestad AJ, Luders T, Esbensen Y, Juul HV, Johansen C, Lyckander LG, Bjornetro T, Inderberg EM, Kersten C, Redalen KR, Ree AH. The mitochondrial DNA constitution shaping T-cell immunity in patients with rectal cancer at high risk of metastatic progression. Clin Transl Oncol. 2022 Jun;24(6):1157-1167. doi: 10.1007/s12094-021-02756-w. Epub 2021 Dec 27. PMID 34961902
- [Derived] Abrahamsson H, Meltzer S, Hagen VN, Johansen C, Bousquet PA, Redalen KR, Ree AH. Sex disparities in vitamin D status and the impact on systemic inflammation and survival in rectal cancer. BMC Cancer. 2021 May 11;21(1):535. doi: 10.1186/s12885-021-08260-2. PMID 33975557
- [Derived] Bakke KM, Meltzer S, Grovik E, Negard A, Holmedal SH, Gjesdal KI, Bjornerud A, Ree AH, Redalen KR. Sex Differences and Tumor Blood Flow from Dynamic Susceptibility Contrast MRI Are Associated with Treatment Response after Chemoradiation and Long-term Survival in Rectal Cancer. Radiology. 2020 Nov;297(2):352-360. doi: 10.1148/radiol.2020200287. Epub 2020 Sep 1. PMID 32870132